CLINICAL TRIAL: NCT05131074
Title: Collabree: A Targeted Behavioral Economics-based Remote Intervention to Improve Medication Adherence in Patients With Hypertension
Brief Title: Collabree: A Remote Intervention to Improve the Regularity of Medication Intake
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Anjali Raja Beharelle (Industry)
Collaborators: MediService AG (Unknown)
Responsible Party: Sponsor-Investigator, Anjali Raja Beharelle, Study Sponsor-Investigator, Collabree AG
Organization: Collabree AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COLLABREE-RS
Record Dates: First submitted 2021-11-11; First posted 2021-11-23 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Hypertension; Medication Adherence
Keywords: Digital Health; Behavioral Change
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group A (Experimental): Patients receive the Collabree mobile phone application with a specific set of functions.
  Interventions: Behavioral: Collabree Mobile Phone Application Medication Adherence Booster
- Intervention Group B (Experimental): Patients receive the Collabree mobile phone application with a specific set of functions.
  Interventions: Behavioral: Collabree Mobile Phone Application Medication Adherence Booster (simplified version)
- Control Group (No Intervention): Patients will not receive the Collabree application.

INTERVENTIONS:
Behavioral: Collabree Mobile Phone Application Medication Adherence Booster — Patients take part in a 90-day program to promote medication adherence and a 90-day follow-up through the Collabree application. Patients will receive more information as to the exact functions and use of the mobile phone application when the application is installed on their mobile phone.
  Arms: Intervention Group A
Behavioral: Collabree Mobile Phone Application Medication Adherence Booster (simplified version) — Patients take part in a 90-day program to promote medication adherence and a 90-day follow-up through the Collabree application. Patients will receive more information as to the exact functions and use of the mobile phone application when the application is installed on their mobile phone.
  Arms: Intervention Group B

SUMMARY:
This is a clinical study to improve the regularity of medication intake for high blood pressure. Adult women and men who are over 50 years old, who have received a prescription drug for high blood pressure from MediService, and who have to take at least 4 tablets per day (of which at least 1 dose of medication per day is for high blood pressure) can participate in this study.

The investigators intend to examine whether Collabree, a mobile phone application, is effective in supporting patients with hypertension to more successfully following their therapy plan in order to improve the regularity of medication intake.

The study includes a 90-day intervention phase and a 90-day follow-up. The study does not require any therapy adjustments and no visits to a study center are necessary. The participants conduct the study independently at home. Participants will also fill out questionnaires.

Participants are randomly assigned to one of 3 groups in a ratio of 1: 1: 1. Two of these groups will receive the Collabree mobile phone application.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent as documented by signature.
2. Over 50 years of age on date of randomization.
3. Patient received prescription medicine against hypertension by post from MediService.
4. Prescribed a therapy against hypertension consisting of 4 or more tablets taken per day. At least 1 dose of medication per day must be against hypertension.
5. Participant administers their own medications.
6. Participant owns a smartphone with a data plan or constant internet access during the study reporting events and at home to use the application.
7. Minimal required smartphone operating system is iOS 12 and Android 8 (Oreo).
8. Adequate communication in German or Swiss-German (all study documentation will only be set to the German language).

Exclusion Criteria:

1. Inability to operate a mobile phone and the Collabree application.
2. Inability to follow the procedures of the study, e.g., due to language problems, psychological disorders, dementia, etc.
3. Enrollment of the Sponsor-Investigator, their family members, employees, and other dependent persons.
4. Participation in another interventional clinical trial.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence | 90 days
  Difference between intervention Group A and the control group in mean medication adherence at endpoint (i.e. the endpoint visit at 90 days) as measured by pill count.

SECONDARY OUTCOMES:
Medication adherence (3 group comparison) | 90 days
  Mean change from baseline in medication adherence (monitored by pill count) at endpoint for the intervention Group A vs. intervention Group B relative to the control group.
Self-reported medication adherence | 90 days
  Mean change from baseline in in-app medication adherence (defined as the number of medications self-reported as "taken" during the intervention period of 90 days divided by the number of prescribed medications listed in the in-app medication plan in that same time period) at endpoint for the intervention Group A vs. intervention Group B relative to the control group.
Self-assessed medication adherence | 90 days
  Mean change from baseline in the score on the Hill-Bone Scale (German version) questionnaire on medication adherence for the intervention Group A vs. intervention Group B relative to the control group at endpoint. The Hill-Bone Compliance to Blood Pressure Therapy Scale (German) scores can range from 14 to 56. A higher score means worse compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Raja Beharelle, PhD, Principal Investigator — Collabree AG
Locations (1):
- Collabree AG, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided